CLINICAL TRIAL: NCT03929900
Title: KoreaN Cohort Study for Outcome in Patients With Chronic Kidney Disease: A Longitudinal Cohort Study of the Chronic Kidney Disease (KNOW-CKD), Phase II Study
Brief Title: KNOW-CKD Cohort, Phase II Study
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kook-Hwan Oh, Professor, Seoul National University Hospital
Other Study IDs: KNOW-CKD2
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Renal progression; Mortality; Complications; Risk factors
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, plasma, random urine will be collected at pre-specified interval
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of KNOW-CKD (KoreaN cohort study for Outcome in patients With Chronic Kidney Disease) study are 1) to establish a CKD cohort representing Korean CKD population for up to 10-year follow-up, and 2) to investigate the renal progression, mortality, complications, risk factors, role of biochemical parameters and the genetic influence. KNOW-CKD Phase I has enrolled 2,238 patients and these patients were divided into four major subgroups depending on the specific causes of CKD : glomerulonephritis, diabetic nephropathy, hypertensive nephropathy, and polycystic kidney disease. In progress, renal progression, complications, and cardiovascular disease of these patients are followed up now.

Since there was a lack of information related to patients' lifestyle, it is necessary to conduct various studies that can be applied to actual clinical status through evaluation of nutrition, cognitive functions, and lifestyles of patients with CKD in South Korea. In addition, researches for high risk patients including diabetic nephropathy, advanced CKD and elderly patients are needed. Thus, KNOW-CKD phase II will enroll the CKD subjects at a more advanced-stage, and older patients than KNOW-CKD phase I subjects.

KNOW-CKD phase II Investigator Group comprises nephrologists, epidemiologists and statisticians from multi-centers in South Korea. KNOW-CKD phase II will enroll 1,500 individuals with estimated glomerular filtration rate between 20 and 60mL/min/1.73m2 (CKD-EPI[Cr] equation) between 2019 and 2021 and follow them until 2016 (for 5~7 years). Unlike phase I, patients diagnosed with glomerulonephritis and ADPKD will be excluded in Phase II.

DETAILED DESCRIPTION:
At enrollment and at pre-specified intervals, laboratory tests will be conducted on the kidney function, biochemical profiles, and anemia. Nutritional evaluation through skin fold, hand grip test, bioelectrical impedence analysis, and 7-point subjective global assessment (SGA), food frequency questionnaire (FFQ) will be conducted in a subgroup of patients. Information on the medical history, health questionnaires, QOL, K-MoCA will also be collected. Web-based case-report forms (CRF) will be used for the systematic management of the patient data.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-79 years
* Estimated glomerular filtration rate 20-60mL/min/1.73m2 based on CKD-EPI(Cr) equation
* Non-dialysis dependent (NDD)

Exclusion Criteria:

* Autosomal dominant polycystic kidney disease
* Unable or unwilling to give consent
* Previously received chronic dialysis
* Previous any organ transplant
* Patients who diagnosed heart failure with NYHA class 3 or 4
* Known liver cirrhosis (Child-pugh class 2 or 3)
* Pregnant women
* Single kidney due to trauma or donation
* Patients who received immunosuppressive agent within the past 1 year
* Patients who diagnosed with glomerulonephritis through kidney biopsy

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-dialysis-dependent, advanced CKD stage between 45 -79 years
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 5 years
  all-cause death, cardiovascular death

SECONDARY OUTCOMES:
Cardiovascular event | 5 years
  major cardiovascular event (MACE)
Renal replacement therapy | 5 years
  end-stage renal disease : dialysis or kidney transplantation
Doubling of serum creatinine or eGFR halving | 5 years
  Doubling of serum creatinine or eGFR halving

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No